CLINICAL TRIAL: NCT02749539
Title: Investigating the Effect of Kinesio Tape Over the Conventional Physical Therapy Management of Shoulder Related Complications in Post-mastectomy Peri-menopausal Females: A Randomized Control Trial
Brief Title: Post Mastectomy Shoulder Problems and Kinesio Taping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dr. Sayed A Tantawy, Associate Professor of Physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/001249
Record Dates: First submitted 2016-04-17; First posted 2016-04-25 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Post Mastectomy Complications
Keywords: Mastectomy; Shoulder Pain; ROM; Kinesio Tape
MeSH Terms: conditions — Shoulder Pain | interventions — Athletic Tape; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Kinesio tape (Experimental): The first 3 kinesio tape application was inhibition technique for supraspinatus, deltoid and teres minor muscles. the fourth Kinesio tape was mechanical correction for the shoulder joint. in addition to active-assistive range of motion exercises (AAROME), active stretching exercises and strengthening exercises for the shoulder joint. Likewise, patients also received postural correction exercises
  Interventions: Device: Kinesio tape; Procedure: physiotherapy program
- Physiotherapy program (Active Comparator): active-assistive range of motion exercises (AAROME), active stretching exercises and strengthening exercises for the shoulder joint. Likewise, patients also received postural correction exercises
  Interventions: Procedure: physiotherapy program

INTERVENTIONS:
Device: Kinesio tape — Standard 2 -inches ( 5-m) Kinesio TexR tape was used for application in the experimental group
  Other Names: Kinesio TexR tape
  Arms: Kinesio tape
Procedure: physiotherapy program — active-assistive range of motion exercises (AAROME), active stretching exercises and strengthening exercises for the shoulder joint. Likewise, patients also received postural correction exercises
  Other Names: exercises

SUMMARY:
Applications of new treatment modality which is Kinesio tape in post mastectomy shoulder problems.

DETAILED DESCRIPTION:
Post-mastectomy complications are often noted and complaints by breast cancer survivors. It often involves the development of chronic arm pain with accompanying limitation of shoulder motion. Aim of the study was to investigate the effect of the kinesio tape (KT) on the shoulder pain and range of motion (ROM).

Method: 74 female patients underwent modified radical mastectomy were involved in this study. They were randomly divided into two groups, experimental who received KT for shoulder joint in addition to conventional physiotherapy program while, the control group received the physiotherapy program only. Outcome measures were visual analogues scale, shoulder ROM and shoulder Pain and Disability Index.

ELIGIBILITY:
Inclusion Criteria:

* Underwent modified radical mastectomy for at least 2 weeks and taking chemotherapy and radiation therapy for stage 1 or II breast cancer.
* Presence of shoulder pain with associated limitation of motion of the shoulder.
* Good compliance and willingness to participate in kinesio taping sessions with a written consent

Exclusion Criteria:

* Still diagnosed with active breast CA at the time of the study.
* Presence of skin hypersensitivity to kinesio tape material.
* Presence of treatment contraindications including the presence of a pacemaker, heart disease, pregnancy, infectious disease, epilepsy thrombophlebitis, arterial hypertension or metastatic cancer .
* Presence of mental disturbances of the sensorium or language problems which can make communication and cooperation problematic.

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2015-02; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 2 weeks change from the baseline scores
  It is a perpendicular line on the scale that corresponded to their perceived pain intensity.

SECONDARY OUTCOMES:
The Shoulder Pain and Disability Index (SPADI) | 2 weeks change from the baseline scores
  It consists of 13 items that assess two domains; a 5-item subscale which measures pain and an 8-item subscale which measures disability. Total score is calculated by averaging the pain and disability subscale scores.

IPD SHARING:
Plan to Share IPD: Yes
publication in a refereed journal